CLINICAL TRIAL: NCT02607280
Title: A JAPANESE, PHASE 3, OPEN-LABEL, 14-WEEK STUDY OF DS-5565 IN PATIENTS WITH PAIN ASSOCIATED WITH DIABETIC PERIPHERAL NEUROPATHY WITH RENAL IMPAIRMENT OR POST-HERPETIC NEURALGIA WITH RENAL IMPAIRMENT
Brief Title: DS-5565 Phase III Study for Renal Impairment in Japanese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS5565-A-J313
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Peripheral Neuropathic Pain; Post-herpetic Neuralgia
Keywords: Diabetic peripheral neuropathic pain; post-herpetic neuralgia; renal impairment
MeSH Terms: conditions — Neuralgia, Postherpetic; Renal Insufficiency | interventions — mirogabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS-5565 group (Experimental): DS-5565 15 mg (for moderate renal impairment) or 7.5 mg (for severe renal impairment), oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Interventions: Drug: DS-5565

INTERVENTIONS:
Drug: DS-5565 — DS-5565 15 mg (for moderate renal impairment) or 7.5 mg (for severe renal impairment), oral administration, Treatment period; 2-weeks titration and 12-weeks fixed dose
  Other Names: mirogabalin

SUMMARY:
Investigate the safety and efficacy of DS-5565 in Japanese subjects with Diabetic Peripheral Neuropathic Pain (DPNP) with renal impairment or Post-Herpetic Neuralgia (PHN) with renal impairment.

DETAILED DESCRIPTION:
The primary objective is the safety and tolerability of DS-5565 in Japanese subjects with moderate to severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* At screening, creatinine clearance (using the Cockcroft-Gault equation): 15-59 mL/min
* At screening, a pain scale of ≥ 40 mm
* Type 1 or type 2 diabetes mellitus at screening (for patients with diabetic peripheral neuropathic pain DPNP only)-. Painful distal symmetric polyneuropathy (for patients with DPNP only)
* post-herpetic neuralgia PHN defined as pain present for more than 3 months after herpes zoster skin rash at screening (for patients with PHN only)

Exclusion Criteria:

* HbA1c (National Glycohemoglobin Standardization Program) > 10.0% (for patients with DPNP only)
* Previous use of neurolytic block (for patients with PHN only)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Baba M, Takatsuna H, Matsui N, Ohwada S. Mirogabalin in Japanese Patients with Renal Impairment and Pain Associated with Diabetic Peripheral Neuropathy or Post-Herpetic Neuralgia: A Phase III, Open-Label, 14-Week Study. J Pain Res. 2020 Jul 17;13:1811-1821. doi: 10.2147/JPR.S255345. eCollection 2020. PMID 32765056

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study from December 2015 to March 2017 at 1 clinic site in Japan.
Groups:
- Moderate Renal Impairment: Participants with moderate RI (creatinine clearance: 30 to 59 mL/min) received DS-5565 2.5 mg BID for the first week and DS-5565 5 mg BID for the second week of the titration period and subsequently received a fixed dose of DS-5565 7.5mg BID for 12 weeks.
- Severe Renal Impairment: Participants with severe RI (creatinine clearance: 15 to 29 mL/min) received DS-5565 2.5 mg QD for the first week and DS-5565 5 mg QD for the second week of the titration period and subsequently received the fixed dose of DS-5565 7.5 mg QD for 12 weeks.
Period: Overall Study
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment
Started | 30 | 5
Received Study Drug | 30 | 5
Completed | 26 | 4
Not Completed | 4 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Decrease in CrCl <15 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 30 | 5 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 27 | 5 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (7.69) | 71.0 (4.06) | 73.4 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 24 | 4 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 5 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 5 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 30 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pain Score (ADPS) at Each Week
Description: Each participant recorded a pain score in the electronic patient diary once daily from the day after the screening visit (Visit 1) to the end of treatment/early termination visit (Visit 10). Prior to taking the study drug each morning, the participant selected the number that best described his or her pain over the past 24 hours on a scale of 0 (no pain) to 10 (worst possible pain). Higher ADPS scores indicated worse outcome. ADPS was the weekly average pain score based on the pain scores from the electronic patient diaries (Pain diary).
  In this outcome, the change from baseline in ADPS is being reported with negative values representing improvements in average daily pain. The larger the negative value (ie. improvement), the greater the improvement in average daily pain.
Time Frame: Baseline to Week 14
Population: ADPS was assessed in the All Enrolled Participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 30 | 5
units on a scale
  Week 1 | -0.14 (0.680) | -0.20 (0.217)
  Week 2 | -0.37 (0.940) | -0.50 (0.937)
  Week 3 | -0.85 (1.294) | -1.83 (1.859)
  Week 4 | -1.13 (1.318) | -2.07 (2.375)
  Week 5 | -0.90 (1.361) | -1.89 (2.278)
  Week 6 | -0.92 (1.285) | -1.82 (1.922)
  Week 7 | -1.22 (1.402) | -1.93 (1.732)
  Week 8 | -1.29 (1.554) | -2.04 (1.735)
  Week 9 | -1.36 (1.540) | -2.21 (1.980)
  Week 10 | -1.33 (1.562) | -2.32 (1.914)
  Week 11 | -1.43 (1.664) | -2.07 (1.584)
  Week 12 | -1.59 (1.636) | -2.10 (1.728)
  Week 13 | -1.84 (1.650) | -2.25 (1.700)
  Week 14 | -1.90 (1.697) | -2.52 (2.026)
Statistical Analysis 1: Comparison: Moderate Renal Impairment; Test type: Other; LS mean change from baseline at Week 14 = -1.79, 95% CI 2-sided [-2.45 to -1.14]
Statistical Analysis 2: Comparison: Severe Renal Impairment; Test type: Other; LS mean change from baseline at Week 14 = -2.07, 95% CI 2-sided [-3.77 to -0.36]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline up to 7 days after last dose, up to 1 year 3 months.
Description: Any adverse event (AE) that emerges on or after first dosing and during the duration of the study treatment (having been absent prior to treatment) or worsens relative to the pre-treatment state.
Arm/Group | Moderate Renal Impairment | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/5
Other Adverse Events (participants affected / at risk) | 17/30 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Renal Impairment (N=30) | Severe Renal Impairment (N=5)
Angina pectoris (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Renal Impairment (N=30) | Severe Renal Impairment (N=5)
Nasopharyngitis (Infections and infestations) | 6 | 2
Somnolence (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 2 | 0
Sensory disturbance (Nervous system disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02607280/Prot_SAP_000.pdf